CLINICAL TRIAL: NCT06574516
Title: The Influence Of Effective Post-Operative Pain Management Following Dental Treatment Under General Anesthesia On Parental Satisfaction And Patient Outcomes
Brief Title: Pain Management Following Dental Treatment Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 448-2021
Record Dates: First submitted 2024-08-25; First posted 2024-08-28 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Pain
Keywords: post operative pain; extraction; general anesthesia
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: blinding of investigators and outcome assessor was possible however no blinding of the participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group 1 (bimodal) (Experimental): participants were given Ibuprofen and Paracetamol alternately every 8 hours for 3 days,
  Interventions: Drug: Ibuprofen 200 mg; Drug: paracetamol
- study group 2 (Experimental): Participants were given Ibuprofen three times daily for 3 days
  Interventions: Drug: Ibuprofen 200 mg
- Control group (Active Comparator): Paracetamol PRN based on parental assessment of pain
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: Ibuprofen 200 mg — Ibuprofen every 8 hours for three days post operatively
  Other Names: Brufen
  Arms: Study group 1 (bimodal); study group 2
Drug: paracetamol — Paracetamol PRN for three days
  Other Names: Panadol
  Arms: Control group; Study group 1 (bimodal)

SUMMARY:
The main goal of this study is to test the efficacy of postoperative pain management for cases undergoing extractions of primary teeth under GA using a validated measure.

Children undergoing extraction of at least one primary molar under general anesthesia GA at King Abdullah University Hospital (KAUH) were randomly assigned into three groups: study group (1) were given Ibuprofen and Paracetamol alternately every 8 hours for 3 days, study group (2) were given Ibuprofen three times daily for 3 days, study group (3) were given Paracetamol prn for 3 days.

pain was assessed using parent's postoperative pain measure (PPPM) on the first, second and third days.

DETAILED DESCRIPTION:
After ensuring the fulfillment of inclusion criteria, data were collected on three phases as follows:

Pre-Operative By interviewing the parents preoperatively during the waiting time, consent was obtained via a consent form , sociodemographic data (name, age, and date of the operation) were also collected using parental questionnaire .

Preoperative pain was measured using WBFPRS. Pre- and postoperative pain scales were explained to parents by the research assistant.

Intra-Operative Data were collected on anesthesia protocol , and dental treatment performed.

Anesthesia Protocol Data about anesthesia protocol were collected to ensure fulfilment of inclusion criteria, this includes mode of induction (IV or inhalational), tube type (nasal or oral), tube size, intra-operative medications (Dexamethasone and analgesia) doses and repetition , cases which did not fulfil the anesthesia protocol were excluded.

Dental Treatment Performed Data on dental procedures were collected including number of extracted teeth, location of extracted teeth (anterior, posterior), and length of dental procedure (in minutes)

Post-Operative Parents were interviewed in the hospital prior to discharge to assess pain 2 hours post operatively using parent's postoperative pain measure (PPPM).

Phone interviews were done to assess postoperative pain using PPPM at home by the same parent at the following intervals: on the night of the procedure, the next day before bed and on the third day before bed. Adherence of parents to pain control prescription was also reported.

ELIGIBILITY:
Inclusion Criteria:

* Fit and healthy patients, ASA I without cognitive or mental disabilities.
* Aged between 4-8 years.
* No preoperative moderate to severe pain.
* Not receiving pain medication prior to GA.
* Not allergic to any of the prescribed medications.
* Undergoing at least one posterior tooth extraction.
* Parent signed the consent form.

Exclusion Criteria:

* Children requiring extraction of permanent molars to ensure standardization.
* Patients who had no extractions at all.
* Cases of difficult intubation as pain of difficult intubation could be confused with dental pain
* Cases where it was necessary to repeat intra-operative analgesic medication (Fentanyl).
* Diclofenac sodium suppository was not given at the end of the procedure.
* Anesthetist did not follow the standardized anesthesia protocol existing in KAUH like cases where a sedative medication like Ketamine was given preoperatively.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2023-04-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of pain control using different medications | 3 days post operative
  Reduction in pain scores using the parental post operative pain measure, by comparing scores immediately post operative with scores on subsequent days. higher scores indicate worse pain

SECONDARY OUTCOMES:
Quality of life of treated children | 2 weeks post operative
  Using Childhood Oral Health Impact Scale (ECOHIS), by comparing pre and postoperative scores, lower scores mean better quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- king Abdulla University Hospital, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No